CLINICAL TRIAL: NCT07274527
Title: The PEARL Trial: A Randomized Trial of Amnioinfusion's Protective Effects on Respiratory and Longitudinal Pediatric Outcomes After Intrapartum Thick Meconium Exposure
Brief Title: Amnioinfusion's Protective Effects on Respiratory and Longitudinal Pediatric Outcomes After Intrapartum Thick Meconium Exposure
Acronym: PEARL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Brock E. Polnaszek MD MPH(c), Assistant Professor and Clinical Investigator, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00054878
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Neonatal Respiratory Distress Related Conditions; Meconium; Perinatal Morbidity; Neonatal Acidosis; Cord Blood; Neonatal Brain Injury; Maternal Morbidity; Mechanical Ventilation; CPAP; Surfactant; Perinatal Death; Amnioinfusion; NICU Admission
Keywords: Amnioinfusion; Meconium; Neonatal morbidity; Developmental Screening; Maternal Morbidity; Neonatal respiratory morbidity; Umbilical cord gas and biomarkers; Healthcare Utilization
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Warm Lactated Ringer Amnioinfusion (Experimental): Standardized warm amnioinfusion consisting of a 500 mL bolus of warmed (37°C) lactated ringer's infused over 30 minutes through an intrauterine pressure catheter (IUPC), followed by a continuous maintenance infusion of 125 mL/hour until the amniotic fluid clears or delivery. Re-administration is permitted if thick meconium persists or the deepest amniotic fluid pocket is <2 cm by ultrasound.
  Interventions: Device: Intrauterine pressure catheter
- Standard of Care (Placebo Comparator): Standard obstetric care will be at the discretion of the delivery provider.
  Interventions: Other: Standard obstetric care at discretion of delivery provider

INTERVENTIONS:
Device: Intrauterine pressure catheter — Standardized warm amnioinfusion consisting of a 500 mL bolus of warmed (37°C) lactated ringer's infused over 30 minutes through an intrauterine pressure catheter (IUPC), followed by a continuous maintenance infusion of 125 mL/hour until the amniotic fluid clears or delivery.
  Other Names: Amnioinfusion
  Arms: Warm Lactated Ringer Amnioinfusion
Other: Standard obstetric care at discretion of delivery provider — Route obstetric care at discretion of delivery provider
  Arms: Standard of Care

SUMMARY:
Thick meconium in the amniotic fluid occurs in about one out of seven pregnancies and increases the chance that a newborn may have breathing problems after birth. These problems can include the need for oxygen, breathing support, admission to the neonatal intensive care unit (NICU), or, in severe cases, meconium aspiration syndrome or persistent pulmonary hypertension.

Although amnioinfusion or placing sterile fluid into the uterus during labor was previously studied as a way to reduce these complications, earlier research had major limitations. Past studies included all types of meconium, used different fluid types and temperatures, had inconsistent protocols, and did not measure biomarkers of inflammation or look at long-term outcomes. As a result, it is still unclear whether a modern, standardized approach to amnioinfusion can meaningfully improve newborn health when the meconium is truly thick.

The PEARL Trial is a randomized clinical trial designed to answer this question. The study will enroll pregnant individuals at or beyond 36 weeks of gestation who develop thick meconium-stained amniotic fluid, confirmed using a simple, objective measurement ("meconium-crit"). Participants will be randomly assigned to receive either:

Warm lactated Ringer's (LR) amnioinfusion through an intrauterine pressure catheter (IUPC), following a standardized protocol, or standard care without amnioinfusion.

The main goal is to determine whether warm LR amnioinfusion reduces short-term breathing problems in newborns. The study also collects umbilical cord blood at birth to evaluate markers of inflammation and potential brain injury, which may help explain why some infants develop complications. Families will also be contacted when their child is 12 months old to complete a developmental questionnaire that is widely used in pediatric practice.

By using a clear definition of thick meconium, a warm LR infusion protocol, fidelity checklists, and long-term follow-up, this trial aims to provide high-quality evidence to guide care in labor and delivery units nationwide.

DETAILED DESCRIPTION:
Thick meconium-stained amniotic fluid is a common intrapartum finding and is associated with increased newborn respiratory morbidity, NICU admission, and long-term developmental concerns. Prior research on amnioinfusion for meconium produced mixed results, largely because earlier trials included all meconium consistencies, used different fluid types and temperatures, did not monitor adherence to infusion protocols, and did not study biologic markers or long-term child outcomes. Because of these limitations, clinicians lack clear evidence about whether modern, standardized amnioinfusion can benefit infants exposed to thick meconium.

The PEARL Trial is designed to address these gaps using a methodologically rigorous, implementation-science-informed approach. The study enrolls maternal-infant dyads at ≥ 36 weeks' gestation with confirmed thick meconium, defined both visually and using an objective "meconium-crit" method that measures the proportion of meconium in the amniotic fluid. After eligibility is confirmed, participants are randomized to receive either a structured warm lactated Ringer's (LR) amnioinfusion protocol or standard obstetric care with no amnioinfusion.

The intervention consists of a 500-mL bolus of warmed LR infused over 30 minutes through an intrauterine pressure catheter, followed by a maintenance infusion until the meconium clears or delivery occurs. Ultrasound checks, infusion parameters, and fluid characteristics are recorded using a fidelity checklist to ensure consistent delivery of the intervention.

The primary outcome is a composite measure of neonatal respiratory morbidity within 72 hours of birth, including need for oxygen, continuous positive airway pressure (CPAP), intubation, inhaled nitric oxide, surfactant therapy, NICU admission, or perinatal death. At birth, umbilical cord blood is collected for gases and for a multiplex panel of inflammatory cytokines and S100B, a biomarker associated with neurologic injury, to better understand biologic pathways linking thick meconium exposure to newborn outcomes. The investigators will also track long-term childhood respiratory morbidity including asthma treatment and severity, reactive airway disease, persistent pulmonary hypertension, bronchopulmonary dysplasia, health care utilization outcomes including but not limited to subspecialty referral, ancillary referrals, emergency room and rehospitalizations.

Long-term follow-up occurs at 12 months corrected age using the Ages and Stages Questionnaire (ASQ-3), a validated tool that screens for communication, motor, problem-solving, and social-emotional development. This allows the trial to explore whether improved intrapartum intervention translates into better developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age greater than or equal to 18 years old
* Singleton pregnancy
* Gestational age of greater than or equal to 36 weeks 0 days gestation
* Cephalic presentation
* Cercial dilation between 2-10 centimeters
* Meconium

Exclusion Criteria:

* Major fetal anomaly
* Multiple gestation
* Eunice Kennedy Shrive National Institute of Child Health and Human Developmet (NICHD) Category III fetal heart tracing
* Contraindication to internal monitors
* Prelabor premature ruptuore of membranes before 36 weeks 0 days gestation, - Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-01-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with composite neonatal respiratory morbidity | 72 hours after delivery
  Composite neonatal respiratory morbidity including continuous positive airway pressure (CPAP) >6 hours, oxygen >24 hours, intubation, persistent pulmonary hypertension (PPHN), surfactant use, inhaled nitric oxide, extracorporeal membrane oxygenation (ECMO), neonatal intensive care unit (NICU) admission, or perinatal death.

SECONDARY OUTCOMES:
Concentration of umbilical cord gas values | At delivery
  Umbilical cord gases including pH, lactate, base excess will be assessed.
Concentration of umbilical cord blood biomarkers | At delivery and if measured in the neonate as a part of usual care
  Human Cytokine/Chemokine Panel A 48-Plex Discovery Assay® (HD48A; Eve Technologies) and other novel markers such as sCD40L, G-CSF, and IFNα2. Additionally, S100B as a validated marker for brain injury will be collected.
Scores on developmental screening | 1 year after delivery
  Predominantly will capture standard developmental screening including the Ages and Stages Questionaires through 1 year of life. Additional information on developmental screening including Sarnat score and referral to subspecialists will be tracked.
Number of participants with composite maternal morbidity | Through 6 weeks postpartum
  Composite morbidity will collect processes related to meconium including postpartum hemorrhage requiring intervention such as estimated blood loss >1000 mililiters (mL) or uterotonics, transexamic acid, blood transfusion or surgical interventions (dilation and curettage, Bakri, Jadha, laparotomy, interventional radiology), endometritis, intraamniotic infection, operative delivery (forceps, vaccum, cesarean), obstetric anal sphincter injury (OASIS), ICU admission, amniotic fluid embolism, and death.

OTHER OUTCOMES:
Number of participants with healthcare utilization | 1 year after delivery
  Capturing all hospitalizatoins, emergency room visits, subspeciality referal, ancillary referrals, and follow-up visits in the first year of life
Number of participants in the Eunice Kennedy Shriver National Institute of Child Health and Human Development Electronic (NICHD) Fetal Monitoring categories | During labor and delivery
  Using standard NICHD data, we will collect and analyze standard electronic fetal monitoring data including things like rates of tachysystole after randomization including categories, declerations, total deceleration area, variablity, accelerations.
Number of participants experiencing pre-defined fidelity metrics | Randomization to 48 hours after birth
  A protocol-specific fidelity checklist will be completed in real time by research staff including Quantification of meconium-crit, Confirmation of cervical dilation ≥ 2 cm, IUPC placement time and verification, Volume and rate of bolus and maintenance infusion, Ultrasound measurements pre- and post-infusion, Fluid color tracking and clearance time, any deviations or complications
Number of participants with neonatal morbidity | 1 year of life
  NICU admission, seizures, hypoxic-ischemic encephalopathy, intracranial hemorrhage and grade, electrolyte abnormalities, hypoglycemia requiring treatment, hyperbilirubinemia requiring phototherapy, neonatal temperature categorized into hypothermia and hyperthermia, suspected and culture proven sepsis, antibiotic administration
Number of participants with placental pathology | Following delivery
  Using contemporary placental pathology recommended and endorse by the College of American Pathologists, we will examine the categories of findings on pathologic examination fo the placenta
Number of participants with composite childhood respiratory morbidity | 1 year of life
  A composite of childhood respiratory morbidity will including tracking for diagnoses realted to respiratory complications such as airway disease, asthma, bronchopulmonary dysplasia, and persistent pulmonary hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital and Medical College of Wisconsin Birth Center, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
IPD data at this time is not a part of our consent process but may be considered on a case-by-case basis with contacting the principal investigator (e.g. a metanalysis) with de-identified data.

REFERENCES:
- [Background] Davis JD, Sanchez-Ramos L, McKinney JA, Lin L, Kaunitz AM. Intrapartum amnioinfusion reduces meconium aspiration syndrome and improves neonatal outcomes in patients with meconium-stained fluid: a systematic review and meta-analysis. Am J Obstet Gynecol. 2023 May;228(5S):S1179-S1191.e19. doi: 10.1016/j.ajog.2022.07.047. Epub 2023 Mar 18. PMID 37164492